CLINICAL TRIAL: NCT05429307
Title: Turkish Adaptation, Validity and Reliability of Exercise Sensitivity Questionnaire
Status: Terminated | Type: Observational
Why Stopped: clinical eligibility for patient recruitment not achieved
Sponsor: Reyhan Kaygusuz (Other)
Responsible Party: Sponsor-Investigator, Reyhan Kaygusuz, Lecturer, Istanbul Demiroglu Bilim University
Organization: Istanbul Demiroglu Bilim University (Other)
Other Study IDs: ESQ
Record Dates: First submitted 2022-06-18; First posted 2022-06-23 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Heart Diseases; Exercise Addiction; Sensitivity
MeSH Terms: conditions — Heart Diseases; Hypersensitivity | interventions — Population

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Population — Turkish Validity and Reliability of The Exercise Sensitivity Questionnair Scale to Turkish society and to make its validity and reliability in Turkish.

SUMMARY:
Interoceptive complex sensations and fear beliefs resulting from cardiac risk factors or cardiovascular disease can further increase one's awareness and attention to bodily situations and cause differences in the interpretation of somatic sensations. These intraceptive somatic sensations may be the underlying factors for participation in exercise and compliance with exercise programs No Turkish questionnaire evaluating unpleasant sensations (Exercise sensitivity) was found. Exercise Sensitivity Questionnaire, which we planned to validate in our study, is a questionnaire developed by Samantha Farris et al. in 2020 to measure anxiety, exercise avoidance behavior and exercise sensitivity, which are frequently observed in individuals with heart disease.

DETAILED DESCRIPTION:
The reliability and validity of the scale will begin with language equivalence and cultural adaptation. The scale will be translated from English to Turkish by two people who are fluent in Turkish and English. A single Turkish translation will be obtained from these two Turkish translations with a common opinion. The scale, which has been translated into Turkish, will be translated into English by two other people who are fluent in Turkish and English. The scale translated into English will be compared with the original. If the developer of the scale, miguel blacutt and Stults-Kolehmainen approves the translation of the scale, participants will be recruited for the study. In the pre-trial phase, a pre- assessment will be conducted with 15 participants to test the intelligibility of the scale. Based on the results of the pre-test phase, the final version of Exercise Sensitivity Questionnaire will be able to be modified. Exercise Sensitivity Questionnaire scale questions and questions in the data collection form face to face 450 participants will be included in the study. In order to evaluate the validity of the Exercise Sensitivity Questionnaire.Tampa Kinesiophobia- Heart and Tampa Kinesiophobia has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 35 years,
* Having a self-reported heart disease (heart failure, acute myocardial infarction, coronary artery disease, coronary by-pass surgery, heart valve surgery, history of stable angina, cardiac have battery)
* To have agreed to participate in the study,
* have internet access,
* Being a mother tongue Turkish.
* Carrying at least two of the cardiac risk factors (hypertension, Type 2 diabetes, hyperlipidemia/dyslipidemia, overweight or obesity (BMI>25), physical inactivity (less than 150 minutes of moderate-intensity exercise per week, smoking)

Exclusion Criteria:

* Not answering all questions
* Cognitive defect or cooperation disorder

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -Population over 35 years of age with self-reported heart disease (heart failure, acute myocardial infarction, coronary artery disease, coronary bypass surgery, heart valve surgery, history of stable angina, pacemaker) voluntarily to participate in the study
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Exercise sensitivity | Beseline
  It is a scale developed by Samantha Farris et al. in 2020 to measure anxiety, exercise avoidance behavior and exercise sensitivity, which are frequently observed in individuals with heart disease. The survey is included in Annex-2. The scale consists of 18 questions in total, consisting of "Not at all", "Very little", "A little", "Too much" and "Too much", and a 5-point Likert type scored between 0-4. Scale scoring is calculated in two subcategories (cardiopulmonary category and pain/weakness category). Scores of questions 6, 8, 11, 12, 13, 14, 15, 15, 16, 17 for the cardiopulmonary category summed and divided by the number of questions. For the pain/weakness category, the scores of questions 1, 2, 3, 4, 5, 6, 7, 9, 10, 18 are added and divided by the number of questions. Higher scores indicate higher sensitivity
Kinesiophobia for Heart Disease | Beseline
  The concept of kinesiophobia was first introduced by Kori et al. Kinesiophobia is also known as fear of movement, avoidance. (Kori et al., 1990). The TAMPA kinesiophobia scale was developed by Vlaeyen et al. (Vlaeyen et al, 2000) to assess the kinesiophobia of patients with low back pain. Bäck et al., on the other hand, rearranged the TAMPA kinesiophobia scale for heart patients and developed the TAMPA Kinesiophobia Rating Scale for the Heart (Bäck et al, 2012). CTSS evaluates the subjective assessment of kinesiophobia in relation to cardiac conditions. The scale consists of four subgroups, which include exercise avoidance, fear of injury, perceived danger for heart problems, and dysfunction. "Strongly disagree" (score It consists of a total of 17 questions on a 4-point Likert scale, scored between 1) and "strongly agree" (score 4).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Demiroglu University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided